CLINICAL TRIAL: NCT02295605
Title: Comparison Between a Land-based and Water-based Muscles Strengthening Program on Patients With Knee Osteoarthritis Randomized Controlled Trial
Brief Title: Comparison Between Land-based and Water-based Exercises for Knee Osteoarthritis: Randomized Controlled Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, André Serra Bley, PhD student, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University of Nove de Julho
Record Dates: First submitted 2014-11-08; First posted 2014-11-20 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Land-based exercises (Experimental): Land-based muscle strengthening exercises protocol
  Interventions: Other: land-based exercises
- Water-based exercises (Experimental): Water-based muscle strengthening exercises protocol
  Interventions: Other: water-based exercises

INTERVENTIONS:
Other: water-based exercises — water-based exercise strengthening protocol for lower limb muscles
  Arms: Water-based exercises
Other: land-based exercises — land-based exercise strengthening protocol for lower limb muscles
  Arms: Land-based exercises

SUMMARY:
Forty six patients with knee osteoarthritis will be randomly allocated into two groups: water-based exercises and land-based exercises. Both of them will receive a strengthening exercise protocol for lower limb muscles. A blind investigator will assess the patients before and immediately after, 3 months and 6 months following the interventions. The main outcomes will be pain, function and strength.

DETAILED DESCRIPTION:
Forty six patients with knee osteoarthritis will be randomly allocated into two groups: water-based exercises and land-based exercises. Both of them will receive a strengthening exercise protocol for lower limb muscles. A blind investigator will assess the patients before and immediately after, 3 months and 6 months following the interventions. The main outcomes will be pain, function, physical performance and strength.

ELIGIBILITY:
Inclusion Criteria:

* Moderate knee osteoarthritis (grade 2 or 3 using the Kellgren-Lawrence radiograph classification), diagnosed based on clinical and radiological criteria of the American College of Rheumatology
* No other lower limb and spine musculoskeletal disorders
* Independent gait
* Body mass index below 32
* Minimum of 4 points in the pain numeric rating scale during climb and descend stairs activities

Exclusion Criteria:

* Cognitive or psychological disorders
* Neurological disorders
* History of post-traumatic knee osteoarthritis
* Knee pain at least 12 months
* Prior surgery of the lower limbs or spine
* Fibromyalgia
* Rheumatoid arthritis
* Cardiovascular disease
* Participating in exercise programs and received treatment for the knee at least 3 months

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-08; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Function | 8 weeks
  Pain and Function scores on the Western Ontario and Mcmaster Universities Osteoarthritis Index (WOMAC questionnaire)

SECONDARY OUTCOMES:
Physical Performance | 8 weeks
  Physical Performance scores on the Timed Up and GO test (TUG)
Strength muscle | 8 weeks
  Strength muscle scores measured by heldheld dynamometer
Lower Limbs Function | 8 weeks
  Function Scores on the Lower Extremity Functional Scale (LEFS)
Pain | 8 weeks
  Pain Scores on the Numeric Pain Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: José Geraldo S Morelli, PhD student, Principal Investigator — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided